CLINICAL TRIAL: NCT02284724
Title: The Effect of Trigger Point Dry Needling to the Multifidus Muscle on Resting and Contracted Thickness of Transversus Abdominis in Subjects With Low Back Pain
Brief Title: Dry Needling to the Multifidus Muscle in Subjects With Low Back Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Nevada, Las Vegas (Other)
Responsible Party: Principal Investigator, Emilio J Puentedura, PT, DPT, PhD, Associate Professor, University of Nevada, Las Vegas
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 1202-4059
Record Dates: First submitted 2014-11-03; First posted 2014-11-06 (Estimated); Last update posted 2018-10-24 (Actual); Status verified 2018-10

CONDITIONS: Low Back Pain, Mechanical
MeSH Terms: conditions — Low Back Pain | interventions — Dry Needling

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Needling (Experimental): Insertion of solid mono-filament needle into lumbar multifidus muscle at both sides of L4/5 segment
  Interventions: Procedure: Dry Needling
- Sham (Other): The plastic tube containing the mono-filament needle will be pressed into the skin over the lumbar multifidus muscle at both sides of L4/5 segment - without insertion through the skin
  Interventions: Procedure: Sham Needling

INTERVENTIONS:
Procedure: Dry Needling
  Arms: Needling
Procedure: Sham Needling
  Arms: Sham

SUMMARY:
To examine for differences in contraction thickness of the transversus abdominis muscle in symptomatic subjects with mechanical lower back pain following the application of dry needling to the lumbar multifidus muscles.

DETAILED DESCRIPTION:
Consenting subjects will be pre-screened for contraindications for dry needling and whether or not they meet the criteria for low back pain. Following acceptance and prior to intervention sessions, subjects will complete a pre-participation questionnaire. This will be used to check for any needle phobia or previous adverse reactions to needling in prospective subjects and analyze potential confounding variables within the subjects participating. Once consented and accepted into the study, subjects will be taught the deep corset contraction (DCC), which is the isolated co-contraction of bilateral transversus abdominis and the deep fibers of lumbar multifidus. Following DCC training, the subject will have a real-time ultrasound transducer applied to the lateral abdominal wall in order to image the three abdominal muscle layers external oblique, internal oblique and transversus abdominis. A relaxed state measure will be taken from the ultrasound image. Subjects will then perform the DCC and a second measure of the abdominal muscles will be taken. A percentage thickness change will be calculated. Prior to treatment, subjects will have been randomly assigned to one of 2 intervention ordered groups: 1) Dry needling: subjects will be placed prone and dry needling to the bilateral multifidus muscles will be performed. Subjects will sense light pressure and their skin will be penetrated by the needle. 2) Sham needling: subjects will be placed prone and the plastic tubes which house the needles for dry needling will be pressed into the bilateral multifidus muscles.Subjects will sense light pressure, but their skin will not be penetrated. All needling and sham needling interventions will be performed under "clean needle" conditions using appropriate skin preparation and use of clean protective gloves by the PI. The needles used will be single-use disposable acupuncture-style needles which come in a plastic tube for easy insertion. Dry needling techniques are techniques that many practicing therapists use for various musculoskeletal conditions, and are also taught by the PI as part of the requirements for the Doctor of Physical Therapy degree. For this study, all needling and sham needling interventions will be performed by the PI who has over 27 years experience in such interventions. Immediately following the needling or sham needling, the real-time ultrasound will be reapplied to measure thickness of the abdominal muscles in the relaxed state and contracted state using the DCC, and percent changes will be calculated. Measurements will be collected by one of three independent researchers who will be blinded to the intervention. An average of 3 measurements will be used to calculate the percent thickness change after the treatment. In addition, the PI performing the needling will remain blinded to ultrasound measurements. Subjects will then be contacted by phone 48 hours as well as one week after the intervention was given in which they will verbally complete questionnaires regarding their degree of pain and level of disability.

ELIGIBILITY:
Inclusion Criteria:

* Age, current symptoms of mechanical low back pain or any symptoms experienced within the last 6 months, and ability to perform DCC.
* Subjects must also report they are comfortable with being 'needled', that is, they should not express a fear of needles and being needled.
* If subjects express fear of needles or being needled, they will be excluded from the study.

Exclusion Criteria:

* History of: abdominal or spinal surgery, significant scoliosis, rheumatoid arthritis, osteoporosis, osteopenia, active ankylosing spondylitis, anticoagulant therapy, hemophilia, lymphedema, and cancer.
* If a subject reports a fear of needles.
* History of adverse reaction to needling (or injection) in the past.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2014-11-01 (Actual); Primary Completion 2018-05-30 (Actual); Study Completion 2018-06-30 (Actual)

PRIMARY OUTCOMES:
Resting thickness transversus abdominis Using real-time ultrasound imaging to measure thickness in milimeters | Immediate
  Using real-time ultrasound imaging to measure thickness in milimeters
Contracted thickness transversus abdominis Using real-time ultrasound imaging to measure thickness in milimeters | Immediate
  Using real-time ultrasound imaging to measure thickness in milimeters

SECONDARY OUTCOMES:
Numeric Pain Rating Scale 10 point pain scale | Immediate and 48 hours later
  10 point pain scale
Oswestry Disability Index | 48 hours later
  Patient reported outcome measure

CONTACTS AND LOCATIONS:
Locations (1):
- University of Nevada Las Vegas - Department of Physical Therapy, Las Vegas, Nevada, United States